CLINICAL TRIAL: NCT06812533
Title: Safety and Efficacy of the Alleviant No-Implant Interatrial Shunt in Patients With Heart Failure and Reduced Ejection Fraction
Brief Title: Alleviant ALLAY-HFrEF Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Alleviant Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIP-0006
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Subjects randomized to the treatment arm will undergo cardiac imaging, femoral vein access and receive the Alleviant ALV1 System device procedure.
  Interventions: Device: Alleviant ALV1 System
- Control (Sham Comparator): Subjects randomized to the control arm will undergo cardiac imaging and sheath placement in femoral vein.
  Interventions: Other: Sham-Control

INTERVENTIONS:
Device: Alleviant ALV1 System — Creation of interatrial shunt
  Arms: Treatment
Other: Sham-Control — Cardiac imaging
  Arms: Control

SUMMARY:
Prospective, multicenter, randomized, sham-controlled, double blind (patient and observer), study designed to evaluate the safety and efficacy of a percutaneously created interatrial shunt using the Alleviant ALV1 System in patients with HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* LVEF ≤ 40%
* NYHA class II, III or ambulatory IV HF
* Receiving optimal, maximally tolerated, stable GDMT

Exclusion Criteria:

* Advanced heart failure
* Life-expectancy < 12 months
* Evidence of right heart dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Composite Primary Endpoint | 12-Month
  The primary endpoint is a composite of all-cause mortality or cardiac transplantation or permanent left ventricular assist device (LVAD) and heart failure events.

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Stone, Principal Investigator — Icahn School of Medicine at Mount Sinai; James Udelson, Principal Investigator — Tufts Medical Center
Locations (43):
- United States (29):
  - Keck Medical Center of USC, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Scripps Clinical Research Services, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Ascension Sacred Heart, Pensacola, Florida
  - Atlanta VA Health Care System, Decatur, Georgia
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Washington University - St Louis, St Louis, Missouri
  - Stony Brook Medicine, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monument Health, Rapid City, South Dakota
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Hendrick Health, Abilene, Texas
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Austin Heart, Austin, Texas
  - NextStage Clinical Research, Waco, Texas
  - Carilion Clinic, Roanoke, Virginia
- Belgium (2):
  - OLV Hospital, Aalst
  - AZ Sint Jan Brugge, Bruges
- Canada (4):
  - Southlake Regional Hospital Centre, Newmarket, Ontario
  - Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Centre Integre Universitaire de Sainte et de Services Scoiiaux de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke (CIUSSS de l'Estrie - CHUS), Montreal, Quebec
  - IUCPQ - Université Laval (Quebec), Québec
- Tbilisi Heart and Vascular, Tbilisi, Georgia
- Uniwesytecki Szpital Kliniczny, Wroclaw, Poland
- Spain (6):
  - Hospital Universitario A Coruna, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital Barcelona, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Valencia Hospital Clinico, Valencia

IPD SHARING:
Plan to Share IPD: No